CLINICAL TRIAL: NCT02706938
Title: Impact of Head of Bed Elevation in Symptoms of Patients With Gastroesophageal Reflux Disease: a Randomized Single-blind Study
Brief Title: Impact of Head of Bed Elevation in Symptoms of Patients With Gastroesophageal Reflux Disease
Acronym: IBELGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IBELGA
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; Head of bed elevation; Quality of life; Nocturnal symptoms; Lifestyle measures
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Randomized single-blind single-centre controlled clinical trial with a 2x2 cross-over design.
Who Masked: Outcomes Assessor
Masking Description: Because HBE is not susceptible to double-blinding, patients allocated to the intervention group will always be aware of the group they belong to. However, the researcher in charge of statistical analysis of data and writing the results report will work with random-generated alphabetical group codes for masking the intervention in each one of the periods of the trial.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Head of bed elevation - Control (Other): Participants will sleep with head of bed raised with standard 20 cm-height wooden blocks during a first period of 6 weeks. After a washout 2 week period, participants will sleep in a bed without inclination for a second period of 6 weeks. During the trial, every patient will receive standard pharmacological treatment with a proton pump inhibitor and/or sodium alginate, according to clinical judgement.
  Interventions: Other: Head of bed elevation; Other: Standard treatment
- Control - Head of bed elevation (Other): Participants will sleep in a bed without inclination during a first period of 6 weeks. After a washout 2 week period, participants will sleep with head of bed raised with standard 20 cm-height wooden blocks for a second period of 6 weeks. During the trial, every patient will receive standard pharmacological treatment with a proton pump inhibitor and/or sodium alginate, according to clinical judgement.
  Interventions: Other: Head of bed elevation; Other: Standard treatment

INTERVENTIONS:
Other: Head of bed elevation — Head of bed elevation will be achieved with a pair of prisms of withered pine tree wood with dimensions (Height x Width x Depth) 20x18x18 cm. Each prism lying on the floor will support one of the head legs of the bed
Other: Standard treatment — Standard pharmacological treatment with a proton pump inhibitor and/or sodium alginate, according to clinical judgement.

SUMMARY:
BACKGROUND: Gastroesophageal reflux disease is a very frequent clinical condition and nocturnal symptoms are a cause of quality of life impairment, poor sleep quality and absenteeism. Head of bed elevation, as a low-cost non pharmacologic anti-reflux treatment is nowadays recommended, but its clinical impact in patients with nocturnal symptoms remains unknown due to inconsistent results and methodological limitations among different clinical trials, most of which were performed before the widespread use of proton pump inhibitors in clinical practice.

HYPOTHESIS: Head of bed elevation is a useful treatment for patients with gastroesophageal reflux disease and nocturnal symptoms, and has a positive impact in quality of life in these patients.

STUDY OBJECTIVE: To assess the effectiveness of head of bed elevation for treatment of patients with gastroesophageal reflux disease and nocturnal symptoms, and to determine the impact of this intervention in quality of life of these patients.

METHODS: Randomized single-blind single-centre controlled clinical trial with a 2x2 cross-over design. A sample of 42 patients attending to the outpatient gastroenterology unit at Clínica Fundadores in Bogotá city, who met the inclusion criteria and had no exclusion criteria were selected to participate. Included patients were randomized to raise the head of bed with standard 20 cm-height wooden blocks or to sleep without bed inclination during the first 6 week period. After a 2 week washout period, allocation was crossed and participants were followed again during a second 6 week period. During the trial, every patient received standard pharmacological treatment with a proton pump inhibitor and/or sodium alginate. After allocation concealment, the researchers in charge of statistical analysis and reporting results were blinded for the non pharmacological intervention under study. Primary outcome was a significant symptom change according to Reflux Disease Questionnaire (RDQ) validated form. Secondary outcomes include impact on quality of life according to Short Form 36 (SF-36) validated questionnaire, patient preference and adverse events of non-pharmacological intervention. Statistical analysis was carried out with STATA 13.0 (Special Edition) for Windows. Differences with a p<0,05 were accepted as statistically significant.

DETAILED DESCRIPTION:
PROBLEM STATEMENT

Gastroesophageal reflux disease (GERD) is a clinical condition characterized by troublesome symptoms and medical complications as a result of reflux of gastric contents into the esophagus. GERD is diagnosed in 4% of primary care outpatient visits and the disease prevalence in Latin-America reaches 12-31%. Nocturnal symptoms have been found in 74% of patients with GERD and are a cause of significant quality of life impairment, when compared with general population and patients with GERD and daytime-only symptoms. Sleep interference secondary to nocturnal retrosternal burning has been associated to lower work productivity, even in patients being treated with proton pump inhibitors (PPI). Due to several physiological factors such as lack of conscious perception of symptoms, reduced salivation and a lower frequency of nocturnal swallowing, a significantly longer acid exposure overnight has been associated to the emergence of complications like esophagitis, more extra-esophageal symptoms and other illnesses such as asthma.

As a low-cost non pharmacological anti-reflux treatment for GERD, head of bed elevation (HBE) is nowadays a moderate-strength recommendation with low level of evidence. Clinical impact of this measure in patients with night-time symptoms remains unknown, due to inconsistent results and methodological limitations among different clinical trials; most of which were performed before the widespread use of proton pump inhibitors in clinical practice. Evidence from several non-randomized studies suggest that HBE could reduce esophageal acid exposure time and could decrease GERD symptoms; however, another study found no significant differences in those same outcomes. On the other hand, all randomized controlled clinical trials published this far show inconsistent results. A study published before widely accepted clinical use of PPI, revealed significant clinical and endoscopic improvement with HBE in patients with GERD and grade C-D esophagitis, when compared to controls. In contrast, a multi-centre clinical trial found no difference in symptom score or antacid use among groups allocated to HBE and control group. All cited studies have methodological limitations and heterogeneity in outcome assessments, which makes difficult conducting a meta-analysis with these data. No published studies evaluating impact of HBE in quality of life or work productivity were found.

SAMPLE SIZE CALCULATION

Sample size was estimated based on the hypothesis that HBE would produce a difference of at least 10% in RDQ and SF-36 scores. Effect size (Cohen d) was calculated as 0,49, keeping in mind an RDQ mean and standard deviation of 3,3±1,0 previously found in Spanish population with symptomatic GERD. An SF-36 mean and standard deviation of 56,9±20,3 reported in Italian population in medical therapy with PPI were also taken into account. The minimally important difference selection was chosen based on the assumption that any difference smaller than 10% would have no clinical relevance. Based on this data, 14 patients per group would yield a power greater than 80% for detection of a minimally important difference as large as or larger than 0,6 points in RDQ questionnaire (range: 1 to 6) and 10 points in SF-36 questionnaire (range: 0 to 100), when using a paired t test. For a complementary analysis of this trial, by using a McNemar test, effect size was recalculated based on published clinical trial data from pre-omeprazole era, according to which 58,8% and 28,6% of patients assigned to placebo improved gastroesophageal reflux symptoms with and without 20 cm HBE, respectively. Based on this data, and maintaining a statistical power of 80%, required sample size was adjusted to a total of 34 patients. G*Power 3.1.9.2 software (Universität Düsseldorf, Düsseldorf, Germany). Finally, estimated sample size was incremented by 20% to avoid that eventual losses of follow-up may alter study power. Therefore, final sample size was 42 patients, 21 patients per group.

DESIGN AND CARVING OF WOODEN PRISMS

84 prisms of withered pine tree wood with dimensions 20x18x18 cm were carved from 9 logs of 300x20x20 cm at Aserrío San Ignacio Ltda. production plant, located in Soacha, Cundinamarca. Given it is an industrial process of chainsaw cutting and wood planing, a quality control was implemented consisting of verification of prism stability while lying on the floor, and the mean height in millimeters of every prism will also be measured and registered. Unsteady products or those with atypical mean heights, defined as a height either exceeding percentile 75 + 1,5 times interquartile range or below percentile 25 - 1,5 times interquartile range, will be discarded and not used during the study. After exclusion of defective prisms,42 groups of wooden prism pairs according to mean height in millimeters were formed and every group was given a random digit generated by computer. Afterwards, every random digit of prism groups was sequentially assigned to a consecutive HBE-allocated patient number, in such a way that every consecutive patient number (among those allocated to HBE) will be linked randomly to a preset known prism height. This additional randomization procedure involving prisms according to their mean height, is planned due to the impossibility to guarantee that prism height will be identical with a precision of ±1 mm, keeping in mind that products will be cut with chainsaw and will be planed as part of an industrial process. After quality control process, mean prism height was found to be a non-normal distributed variable (W:0,908; critic W: 0,979; p: 0,000000), and after applying predetermined exclusion rules for atypical data, 2 pairs of wooden prisms were discarded.

RANDOMIZATION

A random binomial number list (zeroes and ones) will be generated with the statistical software STATA SE 13.0 for Windows and the list will be used for allocation of 42 patients between intervention and control groups in a 1:1 proportion. Each one of the 42 pairs of wooden prisms will be marked with a consecutive number coming from an HBE-allocated patient and the prisms will be stored keeping the marked number out of reach from the sight of the researcher in charge of patient recruiting.

Patients that meet the inclusion criteria, have no exclusion criteria and who give written informed consent, will be assigned a consecutive number during their outpatient visit according to their order of inclusion in the trial. These participants will be randomized to either HBE or control group in the moment that a member of the research team verifies, among the stored prisms, the existence of a prism pair marked with the same number as the consecutive number assigned to the patient. In the case that this pair does exist, then the patient will take home that pair of wooden prisms and use them during the first period of the trial according to spoken and written instructions to be given at that moment. On the contrary, if a pair of wooden prisms marked with the same consecutive number as the patient, does not exist, then it will be understood that the study participant has been allocated to control group during the first period of the trial. The member of the research team who verifies the storehouse of wooden prisms will not be in charge of confirming inclusion and exclusion criteria and will not assign consecutive numbers to patients during outpatient visits.

ALLOCATION CONCEALMENT

The researcher in charge of confirming inclusion and exclusion criteria, fulfilling the Basic Data Formulary and providing the patient with the Informed Consent Format, will not be aware of the allocation sequence order until these 3 documents have been applied to the participant and a consecutive number has been generated according to their order of inclusion in the trial. After that, a member of the research team in the prism storehouse will verify the existence of a prism pair marked with the same number as the consecutive number assigned to the patient, and only in that point allocation status of the participant will be known.

CROSS-OVER

After allocation has been completed, patients in the intervention group will receive a pair of numbered wooden prisms with dimensions 20x18x18 cm along with written instructions about the correct use of the intervention. The patient must sleep with HBE during 6 weeks and both RDQ and SF-36 questionnaires will be applied again at the end of this first period while the participant is still sleeping with HBE. Afterwards, a washout 2 week period follows in which the participant sleeping with HBE will stop using it and will return the pair of wooden prisms to the researchers. After washout period has ended and both RDQ and SF-36 questionnaires have been applied again, patients allocated to the control group during the first period of the study will receive a random pair of prisms and will be instructed to use the prisms for sleeping with HBE during a second period of 6 weeks. Meanwhile, participants initially allocated to the HBE group will be followed as a control group in this second period of the study.

FOLLOW-UP

After participant allocation, telephonic follow up will be made during both periods of the trial with a frequency that is dependent on the intervention group of the patient in that period. Participants in the HBE group will be called weekly for 2 weeks, and then will be called biweekly for a month, until each period of 6 weeks has ended. In contrast, patients in the control group will be called every three weeks along each period. With the purpose of verifying both HBE adherence and correct use of wooden prisms, every participant will be asked to send a photograph of the bed head legs during the follow-up telephone call. The photograph will be received by the researcher via e-mail or smart-phone and will be encoded and saved in a hard disk. At the end of the first period, RDQ and SF-36 questionnaires will be applied and researchers will store the returned prisms during washout period. When washout period has ended, RDQ and SF-36 questionnaires will be applied again in order to be sure of the absence of any carry-over effect in the group initially allocated to HBE. Finally at week 14, RDQ, SF-36 and Patient Preference questionnaires will be administered to complete study ending outcome assessments.

STATISTIC ANALYSIS PLAN

Quantitative and qualitative variables collected with Basic Data Format, RDQ, SF-36 and Patient Preference questionnaires will be typed in a Microsoft Excel 2007 database. Intervention groups will be masked with an alphabetical code provided by an independent collaborator who will not be involved with data analysis or report writing. For statistical processing, database will be imported into STATA SE 13.0 for Windows and descriptive statistics will be generated for each variable. Statistically significant differences will be searched for categorical data using the Chi-square test and normality will be tested for numerical continuous variables using the Shapiro-Wilk test. For normally distributed continuous variables, statistically significant differences will be searched for by using unpaired Student's t test. Alternatively, for not normally distributed variables a Wilcoxon signed rank test will be applied. For complementary processing of primary outcome and secondary outcome quality of life, score difference between periods will be transformed into a binomial variable and a McNemar test will be applied. Differences with one-tail p<0,05 will be accepted as statistically significant. Subgroup analysis will explore differences stratified according to age group, sex, ethnic group, BMI, comorbidities, cups of coffee per day, pharmacological adherence, and length and severity of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal erosions
* Retrosternal pyrosis lasting ≥ 3 months
* Pyrosis and/or regurgitation with a frequency ≥ 3 nights per week
* GERD-associated sleep disturbance (insomnia, poor sleep quality) lasting ≥ 1 month
* GERD-associated sleep disturbance (insomnia, poor sleep quality) with a frequency ≥ 3 nights per week

Exclusion Criteria:

* Non-erosive gastroesophageal reflux disease (NERD)
* Peptic ulcer
* History of upper gastrointestinal surgery (except for cholecystectomy)
* Lactating or pregnant women
* Nighttime shift workers (12 am to 6 am)
* Obstructive sleep apnea hypopnea syndrome
* Chronic obstructive pulmonary disease
* Patients with nocturnal supplementary oxygen requirement
* Orthopnea
* Restless legs syndrome
* Patients consuming more than 3 cups of coffee per day
* Patients planning to travel beyond 3 time zones during study
* Patients being treated with sleep medication (e.g. anxiolytics, antihistamines, benzodiazepines) for less than 3 months
* Patients being treated with sleep medication (e.g. anxiolytics, antihistamines, benzodiazepines), when suspension or dose modification of this drugs is being planned during the study course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan M Villamil Morales, MD, Principal Investigator — Universidad Nacional de Colombia; William A Otero Regino, MD, MSc, Study Director — Universidad Nacional de Colombia, Clínica Fundadores
Locations (1):
- Clínica Fundadores, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Vakil N, Malfertheiner P, Salis G, Flook N, Hongo M. An international primary care survey of GERD terminology and guidelines. Dig Dis. 2008;26(3):231-6. doi: 10.1159/000121352. Epub 2008 May 6. PMID 18463441
- [Background] Salis G. [Systematic review: Epidemiology of gastroesophageal reflux disease in Latin America]. Acta Gastroenterol Latinoam. 2011 Mar;41(1):60-9. Spanish. PMID 21539070
- [Background] Farup C, Kleinman L, Sloan S, Ganoczy D, Chee E, Lee C, Revicki D. The impact of nocturnal symptoms associated with gastroesophageal reflux disease on health-related quality of life. Arch Intern Med. 2001 Jan 8;161(1):45-52. doi: 10.1001/archinte.161.1.45. PMID 11146697
- [Background] Dean BB, Crawley JA, Schmitt CM, Wong J, Ofman JJ. The burden of illness of gastro-oesophageal reflux disease: impact on work productivity. Aliment Pharmacol Ther. 2003 May 15;17(10):1309-17. doi: 10.1046/j.1365-2036.2003.01588.x. PMID 12755844
- [Background] Gross M, Beckenbauer U, Burkowitz J, Walther H, Brueggenjuergen B. Impact of gastro-oesophageal reflux disease on work productivity despite therapy with proton pump inhibitors in Germany. Eur J Med Res. 2010 Mar 30;15(3):124-30. doi: 10.1186/2047-783x-15-3-124. PMID 20452898
- [Background] Orr WC, Heading R, Johnson LF, Kryger M. Review article: sleep and its relationship to gastro-oesophageal reflux. Aliment Pharmacol Ther. 2004 Dec;20 Suppl 9:39-46. doi: 10.1111/j.1365-2036.2004.02239.x. PMID 15527463
- [Background] Orr WC, Allen ML, Robinson M. The pattern of nocturnal and diurnal esophageal acid exposure in the pathogenesis of erosive mucosal damage. Am J Gastroenterol. 1994 Apr;89(4):509-12. PMID 8147351
- [Background] Adachi K, Fujishiro H, Katsube T, Yuki M, Ono M, Kawamura A, Rumi MA, Watanabe M, Kinoshita Y. Predominant nocturnal acid reflux in patients with Los Angeles grade C and D reflux esophagitis. J Gastroenterol Hepatol. 2001 Nov;16(11):1191-6. doi: 10.1046/j.1440-1746.2001.02617.x. PMID 11903734
- [Background] Lopez-Alvarenga JC, Orr W, Vargas-Romero JA, Remes-Troche JM, Morales-Arambula M, Soto-Perez JC, Mateos-Perez G, Sobrino-Cossio S, Teramoto-Matsubara O, Lopez-Colombo A, Orozco-Gamiz A, Saez-Rios A, Arellano-Plancarte A, Chiu-Ugalde J, Tholen A, Horbach S, Lundberg L, Fass R. Relief of Night-time Symptoms Associated With Gastroesophageal Reflux Disease Following 4 Weeks of Treatment With Pantoprazole Magnesium: The Mexican Gastroesophageal Reflux Disease Working Group. J Neurogastroenterol Motil. 2014 Jan;20(1):64-73. doi: 10.5056/jnm.2014.20.1.64. Epub 2013 Dec 30. PMID 24466446
- [Background] Gislason T, Janson C, Vermeire P, Plaschke P, Bjornsson E, Gislason D, Boman G. Respiratory symptoms and nocturnal gastroesophageal reflux: a population-based study of young adults in three European countries. Chest. 2002 Jan;121(1):158-63. doi: 10.1378/chest.121.1.158. PMID 11796445
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Federacao Brasileira de Gastroenterologia; Sociedade Brasileira de Endoscopia Digestiva; Colegio Brasileiro de Cirurgia Digestiva; Sociedade Brasileira de Pneumologia; Associacao Brasileira de Otorrinolaringologia; Cirurgia Cervico-Facial. [Gastroesophageal reflux disease: non-pharmacological treatment]. Rev Assoc Med Bras (1992). 2012 Jan-Feb;58(1):18-24; quiz 25. doi: 10.1590/s0104-42302012000100009. No abstract available. Portuguese. PMID 22392311
- [Background] Dyspepsia and Gastro-Oesophageal Reflux Disease: Investigation and Management of Dyspepsia, Symptoms Suggestive of Gastro-Oesophageal Reflux Disease, or Both. London: National Institute for Health and Care Excellence (NICE); 2014 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK248065/ PMID 25340236
- [Background] Gastroenterological Society of Australia (GESA). Reflux disease: Gastrooesophageal reflux disease in adults. Victoria: GESA 2011. Available from: http://www.gesa.org.au/files/editor_upload/File/Professional/Reflux_Disease.pdf (Accessed Dic, 2014).
- [Background] Stanciu C, Bennett JR. Effects of posture on gastro-oesophageal reflux. Digestion. 1977 Feb;15(2):104-9. doi: 10.1159/000197991. PMID 14044
- [Background] Johnson LF, DeMeester TR. Evaluation of elevation of the head of the bed, bethanechol, and antacid form tablets on gastroesophageal reflux. Dig Dis Sci. 1981 Aug;26(8):673-80. doi: 10.1007/BF01316854. PMID 7261830
- [Background] Khan BA, Sodhi JS, Zargar SA, Javid G, Yattoo GN, Shah A, Gulzar GM, Khan MA. Effect of bed head elevation during sleep in symptomatic patients of nocturnal gastroesophageal reflux. J Gastroenterol Hepatol. 2012 Jun;27(6):1078-82. doi: 10.1111/j.1440-1746.2011.06968.x. PMID 22098332
- [Background] Hamilton JW, Boisen RJ, Yamamoto DT, Wagner JL, Reichelderfer M. Sleeping on a wedge diminishes exposure of the esophagus to refluxed acid. Dig Dis Sci. 1988 May;33(5):518-22. doi: 10.1007/BF01798350. PMID 3359906
- [Background] Harvey RF, Gordon PC, Hadley N, Long DE, Gill TR, Macpherson RI, Beats BC, Tottle AJ. Effects of sleeping with the bed-head raised and of ranitidine in patients with severe peptic oesophagitis. Lancet. 1987 Nov 21;2(8569):1200-3. doi: 10.1016/s0140-6736(87)91332-8. PMID 2890820
- [Background] Pollmann H, Zillessen E, Pohl J, Rosemeyer D, Abucar A, Armbrecht U, Bornhofen B, Herz R. [Effect of elevated head position in bed in therapy of gastroesophageal reflux]. Z Gastroenterol. 1996 Jun;34 Suppl 2:93-9. German. PMID 8767437
- [Background] Kaltenbach T, Crockett S, Gerson LB. Are lifestyle measures effective in patients with gastroesophageal reflux disease? An evidence-based approach. Arch Intern Med. 2006 May 8;166(9):965-71. doi: 10.1001/archinte.166.9.965. PMID 16682569
- [Background] Gerson LB, Fass R. A systematic review of the definitions, prevalence, and response to treatment of nocturnal gastroesophageal reflux disease. Clin Gastroenterol Hepatol. 2009 Apr;7(4):372-8; quiz 367. doi: 10.1016/j.cgh.2008.11.021. Epub 2008 Dec 3. PMID 19111949
- [Background] Nuevo J, Tafalla M, Zapardiel J. [Validation of the Reflux Disease Questionnaire (RDQ) and Gastrointestinal Impact Scale (GIS) in patients with gastroesophageal reflux disease in the Spanish population]. Gastroenterol Hepatol. 2009 Apr;32(4):264-73. doi: 10.1016/j.gastrohep.2008.12.004. Epub 2009 Apr 16. Spanish. PMID 19371971
- [Background] Rossetti G, Limongelli P, Cimmino M, Napoletano D, Bondanese MC, Romano G, Pratilas M, Guerriero L, Orlando F, Conzo G, Amato B, Docimo G, Tolone S, Brusciano L, Docimo L, Fei L. Outcome of medical and surgical therapy of GERD: predictive role of quality of life scores and instrumental evaluation. Int J Surg. 2014;12 Suppl 1:S112-6. doi: 10.1016/j.ijsu.2014.05.034. Epub 2014 Jun 2. PMID 24946311
- [Background] Uniform requirements for manuscripts submitted to biomedical journals: Writing and editing for biomedical publication. J Pharmacol Pharmacother. 2010 Jan;1(1):42-58. No abstract available. PMID 21808590
- [Derived] Villamil Morales IM, Gallego Ospina DM, Otero Regino WA. Impact of head of bed elevation in symptoms of patients with gastroesophageal reflux disease: a randomized single-blind study (IBELGA). Gastroenterol Hepatol. 2020 Jun-Jul;43(6):310-321. doi: 10.1016/j.gastrohep.2020.01.007. Epub 2020 Mar 27. English, Spanish. PMID 32229033
- Available data/document: Study Protocol: Clinical Trial Protocol — https://drive.google.com/open?id=0B6Uam9x9PtiiV2xUcDBKU3RHYU0

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at the outpatient visit of the Gastroenterology, Digestive endoscopy and Liver Diseases Unit in Clínica Fundadores, Bogotá, Colombia. A search for eligible patients was also conducted by using a Local Endoscopy Database with a time frame from 2014 to 2016, and patients with esophagitis were contacted by telephone.
Pre-assignment Details: 1082 out of 1147 potentially eligible patients were excluded prior to randomization. 941 patients did not meet the inclusion criteria and 105 patients had at least one exclusion criteria. 36 patients declined their participation before starting the clinical trial.
Period: First Period, 6 Weeks
Arm/Group | Head of Bed Elevation - Control | Control - Head of Bed Elevation
Started | 32 | 33
Completed | 21 | 31
Not Completed | 11 | 2
Not completed — Adverse Event | 8 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Period, 6 Weeks
Arm/Group | Head of Bed Elevation - Control | Control - Head of Bed Elevation
Started | 21 | 31
Completed (Because this is a crossover trial, only 39 patients who completed both interventions were analyzed.) | 21 (Only data from 20 patients were finally analyzed because of missing data.) | 21 (Only data from 19 patients were finally analyzed because of missing data.)
Not Completed | 0 | 10
Not completed — Adverse Event | 0 | 7
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Head of Bed Elevation - Control | Control - Head of Bed Elevation | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: year] | 57 (8.0) | 54 (12.6) | 55.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 9 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 32 | 32 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Los Angeles Classification [Count of Participants; unit: Participants] — Participants were graded according to the extension of endoscopically confirmed mucosal breaks in the esophagus. Letters from A to D were used for grading, with A meaning a smaller mucosal tear, and D meaning a bigger mucosal tear.
  Participants
    Grade A Esophagitis | 23 | 30 | 53
    Grade B Esophagitis | 8 | 3 | 11
    Grade C Esophagitis | 0 | 0 | 0
    Grade D Esophagitis | 1 | 0 | 1
GERD diagnosis [Median (Inter-Quartile Range); unit: Years] — Self reported years since gastroesophageal reflux disease diagnosis
  Years | 5 [3 to 10] | 5 [2 to 10] | 5 [2 to 10]
GERD-associated sleep disturbance [Median (Inter-Quartile Range); unit: Nights per week] | 3.5 [3 to 5] | 4 [3 to 4] | 4 [3 to 5]
Proton pump inhibitor use [Count of Participants; unit: Participants] | 25 | 31 | 56
Omeprazole use [Count of Participants; unit: Participants] | 4 | 6 | 10
Esomeprazole use [Count of Participants; unit: Participants] | 15 | 22 | 37
Lansoprazole use [Count of Participants; unit: Participants] | 6 | 3 | 9
Sodium Alginate use [Count of Participants; unit: Participants] | 7 | 6 | 13
GERD therapy adherence [Count of Participants; unit: Participants] — The values in the table refer to those participants who were considered having "adherence" to their therapy by means of Morinsky-Green-Levine test. Population: Row population differs from the Overall because of missing data
  Participants
    number analyzed (Participants) | 26 | 30 | 56
    (all) | 14 | 18 | 32
OTC antacid use [Count of Participants; unit: Participants] — Over-the-counter antacid use
  Participants | 4 | 6 | 10
Number of pillows [Median (Inter-Quartile Range); unit: pillows] | 2 [1 to 2] | 2 [1 to 2] | 2 [1 to 2]
Sleep medication [Count of Participants; unit: Participants] | 5 | 5 | 10
Nocturia [Median (Inter-Quartile Range); unit: Nights per week] — The need to wake at night one or more times for voiding
  Nights per week | 3.5 [0.5 to 7] | 6 [1 to 7] | 4 [1 to 7]
Cups of coffee [Median (Inter-Quartile Range); unit: cup] — Patients reported the number of cups of coffee they usually drink daily, taking into account a standard cup of 195 mL.
  cup | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2]
Weight [Mean (Standard Deviation); unit: Kilogram] — Self-reported weight Population: This row populattion differs from the overall because of missed data
  Kilogram
    number analyzed (Participants) | 31 | 33 | 64
    (all) | 67.5 (12.7) | 61.8 (9.5) | 64.6 (11.4)
Height [Mean (Standard Deviation); unit: centimeter] — Self-reported height Population: This row populattion differs from the overall because of missed data
  centimeter
    number analyzed (Participants) | 31 | 33 | 64
    (all) | 161.4 (9.6) | 159.4 (5.7) | 160.4 (7.8)
Body Mass Index [Median (Inter-Quartile Range); unit: Kilogram/square meter] — Population: This row populattion differs from the overall because of missed data
  Kilogram/square meter
    number analyzed (Participants) | 31 | 33 | 64
    (all) | 24.5 [22.9 to 27.8] | 24.9 [22.7 to 25.9] | 24.6 [22.8 to 26.8]
Basal RDQ score [Mean (Standard Deviation); unit: Score on a scale] — Participants were graded according to presence and intensity of reflux symptoms. Reflux Disease Questionnaire (RDQ) was used as a scale with a range from 0 to 6 points, being 0 abscence of symptoms, and 6 the worst intensity of reflux symptoms. Population: This row populattion differs from the overall because of missed data
  Score on a scale
    number analyzed (Participants) | 31 | 32 | 63
    (all) | 3.8 (1.01) | 4 (1.08) | 3.9 (1.04)
SF-36 score [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their overall quality of life. Short Form 36 (SF-36) was used as a scale with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: This row populattion differs from the overall because of missed data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 54 (19.9) | 48.8 (21.4) | 51.3 (20.7)
SF-36 Physical Function domain [Median (Inter-Quartile Range); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account their physical performance. Short Form 36 Physical Function Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: This row populattion differs from the overall because of missed data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 65 [45 to 80] | 55 [35 to 80] | 60 [35 to 80]
SF-36 Physical Role domain [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account if they had role limitations due to physical problems. Short Form 36 Physical Role Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: This row populattion differs from the overall because of missed data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 49.2 (45.7) | 32.2 (42.4) | 40.6 (44.5)
SF-36 Bodily Pain domain [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account their bodily pain. Short Form 36 Bodily Pain Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: This row populattion differs from the overall because of missed data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 43.8 (25) | 40.9 (26.5) | 42.3 (25.6)
SF-36 General Health Domain [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account their general health. Short Form 36 General Health Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: Row population differs from the Overall because of missing data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 51.8 (16.5) | 49.5 (18.2) | 50.6 (17.3)
SF-36 Vitality Domain [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account their vitality. Short Form 36 Vitality Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: Row population differs from the Overall because of missing data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 51 (15.8) | 45.5 (20.7) | 48.2 (18.5)
SF-36 Social Function Domain [Median (Inter-Quartile Range); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account their social performance. Short Form 36 Social Function Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: Row population differs from the Overall because of missing data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 67.5 [55 to 90] | 67.5 [42.5 to 87.5] | 67.5 [55 to 87.5]
SF-36 Emotional Role domain [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account if they had role limitations due to emotional problems. Short Form 36 Emotional Role Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: Row population differs from the Overall because of missing data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 60 (44.1) | 57 (45.7) | 58.5 (44.6)
SF-36 Mental Health domain [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account their mental health. Short Form 36 Mental Health Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent, being 0 the worst quality of life, and 100 the best quality of life. Population: Row population differs from the Overall because of missing data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 60.8 (18) | 57.9 (22.8) | 59.3 (20.5)
SF-36 Transition domain [Mean (Standard Deviation); unit: scores on a scale] — Participants were graded according to a measure of their quality of life, having into account if they felt a transition of their general health during the previous year. Short Form 36 Transition Domain, a sub-scale of SF-36 was used with a range from 0 to 100 percent. Lower percent values mean that participant believes general health is much worse now than one year ago, and higher percent values mean that participant believes general health is much better now than one year ago. Population: Row population differs from the Overall because of missing data
  scores on a scale
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 45 (19) | 37.9 (22.2) | 41.4 (20.8)
Comorbidities [Median (Inter-Quartile Range); unit: Comorbidity] — Number of other chronic illnesses
  Comorbidity | 1.5 [1 to 2] | 2 [1 to 3] | 2 [1 to 3]
Arterial hypertension [Count of Participants; unit: Participants] — Previous diagnosis of chronic arterial hypertension
  Participants | 6 | 5 | 11
Varicose veins [Count of Participants; unit: Participants] — Previous diagnosis of varicose veins in the legs
  Participants | 3 | 8 | 11
Hypothyroidism [Count of Participants; unit: Participants] — Previous diagnosis of hypothyroidism
  Participants | 4 | 6 | 10
Fibromyalgia [Count of Participants; unit: Participants] — Previous diagnosis of fibromyalgia
  Participants | 5 | 5 | 10
Arthrosis [Count of Participants; unit: Participants] — Previous diagnosis of arthrosis
  Participants | 5 | 4 | 9
Irritable bowel syndrome [Count of Participants; unit: Participants] — Previous diagnosis of irritable bowel syndrome
  Participants | 3 | 5 | 8
Depressive disorder [Count of Participants; unit: Participants] — Previous diagnosis of depressive disorder
  Participants | 2 | 6 | 8
Obesity [Count of Participants; unit: Participants] — Participants with a body mass index of 30 or greater Population: Row population differs from the Overall because of missing data
  Participants
    number analyzed (Participants) | 31 | 33 | 64
    (all) | 6 | 2 | 8
Anxiety disorder [Count of Participants; unit: Participants] — Previous diagnosis of anxiety disorder
  Participants | 3 | 4 | 7
Spondylopathy [Count of Participants; unit: Participants] — Previous diagnosis of any spondylopathy
  Participants | 2 | 2 | 4
Type 2 Diabetes Mellitus [Count of Participants; unit: Participants] — Previous diagnosis of type 2 diabetes mellitus
  Participants | 1 | 2 | 3
Other comorbidities [Count of Participants; unit: Participants] — Previous diagnosis of any other comorbidities
  Participants | 10 | 16 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Reflux Disease Questionnaire Scores Administered at Baseline and 6 Weeks After Each Intervention
Description: Change in Reflux Disease Questionnaire Scores administered at baseline and 6 weeks after each intervention. Range from 0 to 6, with a higher punctuation meaning a worse outcome. Symptom change of ≥ 0,6 points from baseline was considered clinically relevant.
Time Frame: Primary outcome will be assessed at baseline and 6 weeks after starting each period
Population: All patients who received the intervention head of bed elevation were grouped, regardless of the arm of the study they came from. Likewise, all participants of any arm who received control intervention were grouped. Only 39 patients who completed both interventions were analyzed because of the crossover nature of this clinical trial.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Head of Bed Elevation: Participants will sleep with head of bed raised with standard 20 cm-height wooden blocks during a first period of 6 weeks.
  Head of bed elevation: Head of bed elevation will be achieved with a pair of prisms of withered pine tree wood with dimensions (Height x Width x Depth) 20x18x18 cm. Each prism lying on the floor will support one of the head legs of the bed
  Standard treatment: Standard pharmacological treatment with a proton pump inhibitor and/or sodium alginate, according to clinical judgement.
- Control: Participants will sleep in a bed without inclination during a first period of 6 weeks.
  Standard treatment: Standard pharmacological treatment with a proton pump inhibitor and/or sodium alginate, according to clinical judgement.
Arm/Group | Head of Bed Elevation | Control
Number analyzed (Participants) | 39 | 39
scores on a scale | -1.2397 (1.2236) | 0.0869 (1.2562)
Statistical Analysis 1: Comparison: Head of Bed Elevation vs Control; Test type: Other — One tail paired t test; p = 0.0002, t-test, 1 sided — A priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.3267, 95% CI 2-sided [0.6263 to 2.0270], Standard Deviation 2.1604
Statistical Analysis 2: Comparison: Head of Bed Elevation vs Control; Test type: Other — McNemar's chi squared statistic; p = 0.0082, McNemar — A priori threshold for statistical significance was 0.05; Risk Difference (RD) = -0.3590, 95% CI 2-sided [-0.6255 to -0.0924]

2. Secondary Outcome: Change in Quality of Life as Assessed by Short Form 36 Questionnaire, Administered at Baseline and 6 Weeks After Each Intervention
Description: Change in Short Form 36 Scores administered at baseline and 6 weeks after each intervention. Range from 0 to 100, with a higher punctuation meaning a better outcome. Quality of life change of ≥ 10 points from baseline was considered clinically relevant.
Time Frame: Secondary outcome will be assessed at baseline and 6 weeks after starting each period
Population: Patients who received the intervention head of bed elevation were grouped, regardless of the arm of the study they came from. Likewise, all participants of any arm who received control intervention were grouped. For crossover reasons, only 39 patients who completed both interventions were analyzed, and 1 patient was excluded because of missing data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Head of Bed Elevation | Control
Number analyzed (Participants) | 38 | 38
scores on a scale | 6.5992 (19.0268) | -0.3139 (17.6856)
Statistical Analysis 1: Comparison: Head of Bed Elevation vs Control; Test type: Other — One tail paired t test; p = 0.099, t-test, 1 sided — A priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -6.9131, 95% CI 2-sided [-17.5987 to 3.7724], Standard Deviation 32.5093
Statistical Analysis 2: Comparison: Head of Bed Elevation vs Control; Test type: Other — McNemar's chi squared statistic; p = 0.8084, McNemar — A priori threshold for statistical significance was 0.05; Risk Difference (RD) = -0.0263, 95% CI 2-sided [-0.2651 to 0.2125]

3. Secondary Outcome: Patient Preference
Description: Percentage of patients who preferred head of bed elevation after trial ending
Time Frame: Secondary outcome will be assessed 14 weeks after starting the trial
Population: All participants who used both head of bed elevation and control interventions, regardless they did not complete the entire trial or did not retrieve all the questionnaires, were asked for their preference between head of bed elevation or control intervention.
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- All Participants: All participants who used both head of bed elevation and control interventions, regardless they did not complete the entire trial or did not retrieve all the questionnaires.
Arm/Group | All Participants
Number analyzed (Participants) | 57
percent of participants | 63.158 [50.635 to 75.681]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 14 weeks for each participant.
Description: The definition of serious adverse event differs from the clinicaltrials.gov definition. In the present study a serious adverse event was the one that led the patient to the suspension of the therapeutic intervention.
  Adverse event information were collected during six serial and telephonic interviews for each patient enrolled in the study.
Arm/Group | Head of Bed Elevation | Control
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/54
Serious Adverse Events (participants affected / at risk) | 15/63 | 0/54
Other Adverse Events (participants affected / at risk) | 24/63 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Head of Bed Elevation (N=63) | Control (N=54)
Varicose veins pain (Vascular disorders) | 4 (4) | 0 (0) — Lower limbs pain attributed to local venous insufficiency
Bed slipping (Product Issues) | 4 (4) | 0 (0) — Participants reported they slip themselves from the surface of the bed, because of bed inclination.
Cervical pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bed unsteadiness (Product Issues) | 3 (3) | 0 (0) — Patients reported their bed was unstable when using wooden blocks for head of bed elevation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Head of Bed Elevation (N=63) | Control (N=54)
Bed slipping (Product Issues) | 16 (16) | 0 (0) — Participants reported they slip themselves from the surface of the bed, because of bed inclination.
Varicose veins pain (Vascular disorders) | 6 (6) | 0 (0) — Lower limbs pain attributed to local venous insufficiency
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bed unsteadiness (Product Issues) | 1 (1) | 0 (0)
Sexual activity interference (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Patients reported their sexual activity was difficult when using wooden blocks for head of bed elevation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT02706938/Prot_SAP_ICF_000.pdf